CLINICAL TRIAL: NCT04938830
Title: A Phase 3, Multicenter, Randomized, Partially Blinded, Palivizumab- Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of MK-1654 in Infants and Children at Increased Risk for Severe RSV Disease
Brief Title: Clesrovimab (MK-1654) in Infants and Children at Increased Risk for Severe Respiratory Syncytial Virus (RSV) Disease (MK-1654-007)
Acronym: SMART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1654-007; MK-1654-007 (Other: MSD); jRCT2031210664 (Registry Identifier: jRCT); 2022-500752-39-00 (Registry Identifier: EU CT); U1111-1278-0093 (Registry Identifier: UTN); 2020-005996-11 (EudraCT Number)
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — MK-1654; Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clesrovimab (Experimental): Participants will receive intramuscular (IM) injections of clesrovimab and placebo
  Interventions: Biological: Clesrovimab; Biological: Placebo
- Palivizumab (Active Comparator): Participants will receive IM injections.
  Interventions: Biological: Palivizumab

INTERVENTIONS:
Biological: Clesrovimab — IM injection
  Other Names: MK-1654
  Arms: Clesrovimab
Biological: Palivizumab — IM injection
  Arms: Palivizumab
Biological: Placebo — IM injection
  Arms: Clesrovimab

SUMMARY:
This study aims to evaluate the safety and tolerability of clesrovimab compared to palivizumab as assessed by the proportion of participants experiencing adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Participants at increased risk for severe RSV infection recommended to receive palivizumab in accordance with national or local guidelines or professional society recommendations.
* Is available to complete the follow-up period.

Exclusion Criteria:

* Requires mechanical ventilation at time of enrollment.
* Has a life expectancy <6 months.
* Has known hepatic or renal dysfunction, or chronic seizure disorder.
* Is hospitalized at the time of randomization unless discharge is expected within 7 days after randomization.
* Has severe immunodeficiency or is severely immunocompromised.
* Has known hypersensitivity to any component of clesrovimab or palivizumab.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1003 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Participants with solicited injection-site Adverse Events (AEs) in RSV Season 1 | Up to 5 days
  Percentage of participants with solicited injection-site AEs in RSV Season 1
Participants with solicited daily body temperature with fever in RSV Season 1 | Up to 5 days
  Percentage of participants with solicited daily body temperature with fever in RSV Season 1
Participants with solicited systemic AEs in RSV Season 1 | Up to 5 days
  Percentage of participants with solicited systemic AEs in RSV Season 1
Participants with anaphylaxis/hypersensitivity AEs of special interest (AESI) in RSV Season 1 | Up to 42 days
  Percentage of participants with anaphylaxis/hypersensitivity AESI in RSV Season 1
Participants with rash AESI in RSV Season 1 | Up to 42 days
  Percentage of participants with rash AESI in RSV Season 1
Participants with non-serious AEs in RSV Season 1 | Up to 42 days
  Percentage of participants with non-serious AEs in RSV Season 1
Participants with serious AEs (SAEs) through the duration of participation in RSV Season 1 | Up to 365 days
  Percentage of participants with serious AEs (SAEs) through the duration of participation in RSV Season 1

SECONDARY OUTCOMES:
Participants with RSV-associated medically attended lower respiratory infection (MALRI) in RSV Season 1 | Up to 150 days
  Percentage of participants with RSV-associated medically attended lower respiratory infection (MALRI) in RSV Season 1
Participants with RSV-associated hospitalization in RSV Season 1 | Up to 150 days
  Percentage of participants with RSV-associated hospitalization in RSV Season 1
Participants with solicited injection-site AEs in RSV Season 2 | From approximately 393 days up to 400 days
  Percentage of participants with solicited injection-site AEs in RSV Season 2
Participants with solicited daily body temperature with fever in RSV Season 2 | From approximately 393 days up to 400 days
  Percentage of participants with solicited daily body temperature with fever in RSV Season 2
Participants with solicited systemic AEs in RSV Season 2 | From approximately 393 days up to 400 days
  Percentage of participants with solicited systemic AEs in RSV Season 2
Participants with anaphylaxis/hypersensitivity AESI in RSV Season 2 | From approximately 393 days up to 440 days
  Percentage of participants with anaphylaxis/hypersensitivity AESI in RSV Season 2
Participants with rash AESI in RSV Season 2 | From approximately 393 days up to 440 days
  Percentage of participants with rash AESI in RSV Season 2
Participants with non-serious AEs in RSV Season 2 | From approximately 393 days up to 440 days
  Percentage of participants with non-serious AEs in RSV Season 2
Participants with SAEs in RSV Season 2 | From approximately 393 days up to 575 days
  Percentage of participants with SAEs in RSV Season 2
Concentration of clesrovimab in RSV Season 1 | Up to 240 days
  Serum concentration of clesrovimab after dose of clesrovimab in RSV Season 1
Concentration of clesrovimab in RSV Season 2 | From approximately 393 days up to 550 days
  Serum concentration of clesrovimab after dose of clesrovimab in RSV Season 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (146):
- United States (29):
  - Miller Children's & Women's Hospital Long Beach ( Site 0001), Long Beach, California
  - Children's Hospital of Orange County ( Site 0047), Orange, California
  - Children's Hospital Colorado ( Site 0011), Aurora, Colorado
  - Children's National Medical Center ( Site 0020), Washington D.C., District of Columbia
  - Orlando Health - Arnold Palmer Hospital-Orlando Health-Arnold Palmer Hospital Pulmonary and Sleep M ( Site 0022), Orlando, Florida
  - Nemours Children's Health, Lake Nona Medical City ( Site 0032), Orlando, Florida
  - University of South Florida-Department of Pediatrics ( Site 0045), Tampa, Florida
  - Morehouse School Of Medicine ( Site 0049), Atlanta, Georgia
  - Clinical Research Prime ( Site 0046), Idaho Falls, Idaho
  - University of Kentucky HealthCare - Turfland ( Site 0044), Lexington, Kentucky
  - Our Lady of the Lake Children's Hospital ( Site 0031), Baton Rouge, Louisiana
  - Tulane University School of Medicine ( Site 0010), New Orleans, Louisiana
  - M Health Fairview University of Minnesota Masonic Children's Hospital, West Bank-Peds Research ( Site 0037), Minneapolis, Minnesota
  - Rutgers University-Pediatric Clinical Research Center ( Site 0007), New Brunswick, New Jersey
  - NYU Langone Hospital - Long Island-Pediatrics ( Site 0028), Mineola, New York
  - University of Rochester Medical Center ( Site 0017), Rochester, New York
  - The University of North Carolina at Chapel Hill ( Site 0035), Chapel Hill, North Carolina
  - Duke University ( Site 0021), Durham, North Carolina
  - Dayton Children's Hospital ( Site 0053), Dayton, Ohio
  - Tribe Clinical Research, LLC ( Site 0002), Greenville, South Carolina
  - Driscoll Children's Hospital ( Site 0025), Corpus Christi, Texas
  - DHR Health Institute for Research and Development ( Site 0029), Edinburg, Texas
  - Christus Children's-Clinical Research Center ( Site 0038), San Antonio, Texas
  - University Hospital-Pediatrics ( Site 0019), San Antonio, Texas
  - Road Runner Research, Ltd ( Site 0052), San Antonio, Texas
  - Intermountain - Primary Children's Hospital ( Site 0026), Salt Lake City, Utah
  - Multicare Rockwood Main Clinic-Rockwood Pediatrics ( Site 0004), Spokane, Washington
  - Providence Sacred Heart Medical Center & Children's Hospital ( Site 0030), Spokane, Washington
  - MultiCare Health System-Baker Center ( Site 0036), Tacoma, Washington
- Australia (2):
  - Mater Misericordiae Limited-Neonatalogy ( Site 0102), Brisbane, Queensland
  - Telethon Kids Institute-Vaccine Trials Group ( Site 0101), Nedlands, Western Australia
- Canada (3):
  - Alberta Children's Hospital-Department of Pediatrics ( Site 0180), Calgary, Alberta
  - Canadian Center for Vaccinology ( Site 0179), Halifax, Nova Scotia
  - CHU Sainte-Justine ( Site 0178), Montreal, Quebec
- Chile (3):
  - Clínica Alemana de Santiago-Neonatology department ( Site 0207), Santiago, Region M. de Santiago
  - Hospital Roberto del Río-Infectología Pediátrica ( Site 0205), Santiago, Region M. de Santiago
  - Hospital Padre Hurtado-NEONATOLOGY/PEDIATRICS ( Site 0201), Santiago, Region M. de Santiago
- Colombia (5):
  - Fundación Hospitalaria San Vicente de Paúl ( Site 0233), Medellín, Antioquia
  - Clínica Universitaria Bolivariana ( Site 0227), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0235), Barranquilla, Atlántico
  - Sociedad de Cirugía de Bogotá - Hospital de San Jose ( Site 0230), Bogotá, Bogota D.C.
  - Clínica Imbanaco S.A.S ( Site 0229), Cali, Valle del Cauca Department
- Czechia (2):
  - Fakultni nemocnice Ostrava-Oddeleni neonatologie ( Site 0252), Ostrava, Moravskoslezský kraj
  - Institute for the Care of Mother and Child ( Site 0251), Prague, Praha 4
- Finland (6):
  - FVR, Kokkolan rokotetutkimusklinikka ( Site 0304), Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka ( Site 0303), Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka ( Site 0301), Tampere, Pirkanmaa
  - FVR, Seinäjoen rokotetutkimusklinikka ( Site 0305), Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka ( Site 0302), Turku, Southwest Finland
  - MeVac - Meilahti Vaccine Research Center ( Site 0306), Helsinki, Uusimaa
- France (3):
  - Bordeaux University Hospital - Pellegrin-Pediatrics ( Site 0332), Bordeaux, Aquitaine
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de N-Centre de Recherche Clinique Pédiatriq ( Site 0330), Caen, Calvados
  - Centre Hospitalier de Versailles André Mignot-NEONATOLOGY ( Site 0331), Le Chesnay, Yvelines
- Germany (9):
  - Universitaetsklinikum Freiburg ( Site 0365), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg-Zentrum für Kinder-und Jugendmedizin ( Site 0366), Heidelberg, Baden-Wurttemberg
  - Dr. von Haunersches Kinderspital ( Site 0358), Munich, Bavaria
  - München Klinik Harlaching ( Site 0351), Munich, Bavaria
  - Medizinische Hochschule Hannover ( Site 0364), Hanover, Lower Saxony
  - Kinder und Jugendaerztliche Gemeinschaftspraxis Bedikian & Bouikidis ( Site 0359), Oberhausen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Kinder- und Jugendmedizin ( Site 0363), Dresden, Saxony
  - Universitätsklinikum Leipzig-Neonatology ( Site 0354), Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein-Pediatrics ( Site 0361), Lübeck, Schleswig-Holstein
- Greece (4):
  - Aghia Sophia Children's Hospital-First Department of Pediatrics, National and Kapodistrian Universi ( Site 0852), Athens, Attica
  - Children's Hospital Aglaia Kyriakou-2nd Department of Pediatrics NKUA ( Site 0854), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL-3rd Department of Pediatrics ( Site 0855), Chaïdári, Attica
  - Hippokration University Hopsital-3rd Pediatric Department ( Site 0851), Thessaloniki, Central Macedonia
- Hong Kong (2):
  - Prince of Wales Hospital ( Site 0926), Shatin
  - Tuen Mun Hospital ( Site 0927), Tuenmen
- Hungary (8):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház-Újszülött Intenzív Osztály ( Site 0388), Miskolc, Borsod-Abauj Zemplen county
  - Bajai Szent Rókus Kórház ( Site 0386), Baja, Bács-Kiskun county
  - Bacs-Kiskun Megyei Korhaz-Pediatrics ( Site 0380), Kecskemét, Bács-Kiskun county
  - Szabolcs-Szatmar-Bereg Varmegyei Korhazak es Egyetemi Oktatokorhaz - Gyermekosztaly ( Site 0376), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Péterfy Kórház-Rendelőintézet és Manninger Jenő Országos Traumatológiai Intézet-PIC ( Site 0384), Budapest
  - Semmelweis University-Szülészeti és Nőgyógyászati Klinika PIC ( Site 0381), Budapest
  - Gottsegen György Országos Kardiovaszkuláris Intézet ( Site 0383), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0378), Debrecen
- Italy (6):
  - Ospedale Pediatrico Bambino Gesù IRCCS-UOC Broncopneumologia ( Site 0427), Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 0426), Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 0432), Milan, Lombardy
  - ASST Fatebenefratelli Sacco ( Site 0434), Milan, Lombardy
  - Azienda Ospedaliera di Padova-Department of Women and Child Health ( Site 0428), Padua, Veneto
  - Azienda Ospedaliero Universitaria di Parma-UO Clinica Pediatrica ( Site 0433), Parma
- Japan (8):
  - Fukuoka Children's Hospital ( Site 0452), Fukuoka, Fukuoka
  - Iizuka Hospital ( Site 0457), Iizuka, Fukuoka
  - Japan Community Healthcare Organization Kyushu Hospital ( Site 0454), Kitakyushu-shi, Fukuoka
  - Maebashi Red Cross Hospital ( Site 0451), Maebashi, Gunma
  - Ibaraki Children's Hospital ( Site 0458), Mito, Ibaraki
  - Nihon University Itabashi Hospital ( Site 0453), Itabashiku, Tokyo
  - Shizuoka Saiseikai General Hospital ( Site 0456), Shizuoka
  - National Center for Child Health and Development ( Site 0455), Tokyo
- Malaysia (6):
  - Hospital Raja Perempuan Zainab II-Department of Pediatric ( Site 0477), Kota Bharu, Kelantan
  - University Malaya Medical Centre-Department of Paediatrics ( Site 0480), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 0482), George Town, Pulau Pinang
  - Sabah Women and Children Hospital ( Site 0478), Kota Kinabalu, Sabah
  - Hospital Sibu ( Site 0476), Sibu, Sarawak
  - Hospital Tunku Azizah-Paediatric ( Site 0481), Kuala Lumpur
- Mexico (6):
  - Morales Vargas Centro de Investigacion ( Site 0509), León, Guanajuato
  - Centro de Investigación Médico Biológica y Terapia Avanzada ( Site 0502), Guadalajara, Jalisco
  - Instituto Nacional de Pediatria ( Site 0506), Mexico City, Mexico City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C. ( Site 0508), Durango
  - Oaxaca Site Management Organization ( Site 0504), Oaxaca City
  - ONCOLOGICO POTOSINO, S.C. ( Site 0505), San Luis Potosí City
- New Zealand (2):
  - Capital and Coast District Health Board-Clinical Trials Unit ( Site 0527), Newtown, Wellington Region
  - Middlemore Clinical Trials ( Site 0526), Auckland
- Oslo Universitetssykehus Ullevål ( Site 0551), Oslo, Norway
- Peru (2):
  - Instituto Nacional Cardiovascular INCOR Carlos Peschiera Carrillo - EsSalud ( Site 0577), Jesús María, Lima
  - HOSPITAL DOCENTE MADRE-NIÑO SAN BARTOLOME-NEUMOLOGIA PEDIATRICA ( Site 0576), Lima
- UPR Medical Sciences Campus-Pediatrics ( Site 0626), San Juan, Puerto Rico
- KK Women's and Children's Hospital-Department of Neonatology ( Site 0877), Singapore, South West, Singapore
- South Africa (7):
  - Reimed ( Site 0706), Boksburg, Gauteng
  - Chris Hani Baragwanath Academic Hospital ( Site 0701), Soweto, Gauteng
  - King Edward VIII Hospital ( Site 0704), Durban, KwaZulu-Natal
  - Family Clinical Research Unit (Fam-Cru)-Pediatric ( Site 0703), Cape Town, Western Cape
  - Panorama Medical Centre ( Site 0702), Cape Town, Western Cape
  - MRC Unit on Child And Adolescent Health-Department of Paediatrics and child Health ( Site 0710), Cape Town, Western Cape
  - 2 Military Hospital ( Site 0708), Cape Town, Western Cape
- Spain (10):
  - Hospital Germans Trias i Pujol ( Site 0738), Badalona, Barcelona
  - Hospital Sant Joan de Déu ( Site 0730), Esplugues de Llobregat, Barcelona
  - Hospital Universitary General de Catalunya-Pediatrics ( Site 0737), Sant Cugat del Vallès, Barcelona
  - CHUS - Hospital Clinico Universitario-Servicio de Pediatría ( Site 0731), Santiago de Compostela, La Coruna
  - Hospital Universitario HM Monteprincipe-pediatric ( Site 0743), Boadilla del Monte, Madrid
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 0739), Pozuelo de Alarcón, Madrid
  - Hospital Universitario 12 de Octubre-Unidad Pediátrica de Investigación y Ensayos Clínicos ( Site 0728), Madrid, Madrid, Comunidad de
  - Hospital Universitario Central de Asturias ( Site 0740), Oviedo, Principality of Asturias
  - Hospital Universitario La Paz ( Site 0726), Madrid
  - Grupo Pediatrico Uncibay ( Site 0734), Málaga
- Taiwan (4):
  - Taichung Veterans General Hospital ( Site 0754), Taichung
  - National Taiwan University Hospital ( Site 0751), Taipei
  - Mackay Memorial Hospital-Pediatrics ( Site 0753), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0752), Taoyuan District
- Thailand (3):
  - Chulalongkorn University-Pediatrics ( Site 0777), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Pediatric Infectious Diseases ( Site 0778), Bangkok, Bangkok
  - Songklanagarind hospital-Department of Pediatrics ( Site 0776), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (5):
  - cukurova universty ( Site 0805), Sarçam, Adana
  - Ankara University Hospital Cebeci ( Site 0801), Ankara
  - Gazi Universitesi ( Site 0806), Ankara
  - Ankara Bilkent Şehir Hastanesi. ( Site 0807), Ankara
  - Erciyes University Medical Faculty-pediatric infection ( Site 0804), Kayseri
- United Kingdom (8):
  - Whipps Cross University Hospital ( Site 0846), London, England
  - St. George's Hospital ( Site 0845), London, England
  - Queen Elizabeth University Hospital ( Site 0842), Glasgow, Glasgow City
  - Evelina London Children's Hospital ( Site 0829), London, Great Britain
  - Southampton General Hospital ( Site 0826), Southampton, Hampshire
  - Barts Health NHS Trust-Children's Clinical Research Facility ( Site 0844), London, London, City of
  - The John Radcliffe Hospital-Paediatrics Infectious Diseases ( Site 0827), Oxford, Oxfordshire
  - Alder Hey Children's Hospital-Paediatric Respiratory Medicine ( Site 0843), Liverpool

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Zar HJ, Bont LJ, Manzoni P, Munoz FM, Ramilo O, Chen PY, Novoa JM, Ordonez GA, Tsolia M, Tapiero B, Acuna-Avila MI, Castellanos JM, Meyer M, Morioka I, Chen Z, Railkar RA, Zang X, Maas BM, Likos A, Lee AW, Castagnini LA, Sinha A; SMART (MK-1654-007) Study Group. Clesrovimab in Infants and Children at Increased Risk for Severe RSV Disease. N Engl J Med. 2025 Oct 2;393(13):1343-1345. doi: 10.1056/NEJMc2506107. Epub 2025 Sep 17. No abstract available. PMID 40961423
- [Derived] Sinha A, Railkar RA, Castagnini L, Guerra A, Likos A, Lutkiewicz J, Maas BM, Zang X, Roadcap BA, Choi Y, Nahhas GJ, Arriola CS, Bont L, Manzoni P, Ramilo O, Munoz FM, Finelli L, Lee AW. Evaluation of a monoclonal antibody against respiratory syncytial virus, clesrovimab, in infants and children: Comprehensive rationale and study design for the late-stage clinical trials. Contemp Clin Trials. 2025 Oct;157:107995. doi: 10.1016/j.cct.2025.107995. Epub 2025 Jun 30. PMID 40602662
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26175&tenant=MT_MSD_9011